CLINICAL TRIAL: NCT02080572
Title: Parkinstep: Automated PD Gait and Balance Assessment for Optimizing DBS
Status: Completed | Type: Observational
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other); University of Cincinnati (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: AG033947-03A1; 2R44AG033947-03A1 (NIH)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease With Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinson's Disease with DBS: Individuals with Parkinson's disease and deep brain stimulation will be recruited.

SUMMARY:
Changes in deep brain stimulation (DBS) settings can have a delayed effect on gait function, which makes it impractical to optimize DBS for gait parameters in the clinic. Wearable movement sensors could be used to assess gait impairment in the patient's home hours after treatment adjustments are made in the clinic. This study aims to quantitatively evaluate the effects of turning off deep brain stimulation on lower extremity and gait function over three hours. This study will provide vital information about our patient worn system's ability to detect changes in lower impairment over time, which could be used to assist with DBS tuning for the lower extremities and gait in the future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease
* Age > 21
* Underwent DBS surgery targeting the subthalamic nucleus (STN)
* Bilateral or midline involvement when "off" DBS/medication state
* Clinical history of gait impairment or freezing of gait

Exclusion Criteria:

* "Parkinson's plus" syndrome, secondary, or atypical Parkinson's disease
* Underwent DBS surgery targeting the ventral intermediate (VIM)
* Unable to walk independent of a wheelchair (use of assistive devices, like a cane, is okay for this study)
* Dementia (determined by a neuropsychological assessment).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Parkinson's disease, gait impairment, and deep brain stimulation will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Effect of DBS cessation on motor function over time | All data will be collected within a single session not to exceed 4 hours. All data will be analyzed within one month of study completion.
  Motor function evaluations (movement speed and magnitude) will be collected at various time points after DBS cessation. The effects over time will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Giuffrida, PhD, Principal Investigator — Great Lakes NeuroTechnologies
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Case Western, Cleveland, Ohio